CLINICAL TRIAL: NCT05020730
Title: A 12-Week Double-Blind, Placebo-Controlled Randomized Phase 2 Trial With a 12-Week Open-Label Extension to Determine the Immunomodulatory Activity of PTM-001 in Patients With Hidradenitis Suppurativa
Brief Title: Trial to Determine the Immunomodulatory Activity of PTM-001 in Patients With Hidradenitis Suppurativa
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Phoenicis Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTM-001-01
Record Dates: First submitted 2021-08-18; First posted 2021-08-25 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Suppurativa; HS; Inflammatory skin disease; Humira; P2X7; IL-1β
MeSH Terms: conditions — Hidradenitis Suppurativa; Dermatitis

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive PTM-001 (400 mg) or matching placebo every day for 12 weeks after which all patients will receive open-label PTM-001 400 mg daily for an additional 12 weeks
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PTM-001 400 mg daily for 12 weeks (Experimental)
  Interventions: Drug: PTM-001
- Placebo daily for 12 weeks (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PTM-001 — PTM-001 (400 mg) every day for 12 weeks
  Arms: PTM-001 400 mg daily for 12 weeks
Drug: Placebo — Matching placebo every day for 12 weeks
  Arms: Placebo daily for 12 weeks

SUMMARY:
Study PTM-001-01 is a 12-week, randomized, placebo controlled, double blind study with a 12 week open-label extension to examine the immunomodulatory activity of PTM-001 in participants with Hidradenitis Suppurativa (HS). Participants will be randomized to receive PTM-001 (400 mg) or matching placebo every day for 12 weeks after which all participants will receive open-label PTM-001 400 mg daily for an additional 12 weeks. Randomization will be stratified by Hurley Stage.

ELIGIBILITY:
Inclusion Criteria:

* Had onset of symptoms consistent with HS at least 6 months prior to Screening.
* Has had active HS for at least 2 months.
* Has ≥ 5 HS abscesses or inflammatory nodules at Screening.
* Agrees to maintain baseline wound care and antibiotic therapy, including oral antibiotics, for the duration of the trial.
* Agrees to use contraception

Exclusion Criteria:

* Has other skin disease or condition that can interfere with HS assessment.
* Has a positive test for TB, HIV, hepatitis B and/or hepatitis C at Screening.
* Has a history of retinopathy or known clinically significant cardiovascular or hematologic conditions.
* Has taken any biologic drug within 3 serum half-lives. A list of potential biologics and their half-lives
* Has started oral antibiotics within 28 days of Study Day 1.
* Has, within 2 weeks prior to Day 1, received a medication prohibited based on cytochrome P450 (CYP3A4) interaction
* Has such extensive disease that, in the opinion of the Investigator, it is difficult to discriminate between active lesions and scarring.
* Has more than 15 active tunnels at Screening.
* Is pregnant, nursing or considering becoming pregnant.
* Has a history of malignancy except non-melanoma skin cancer or cervical carcinoma in situ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Effect of PTM-001 on IL-1β protein levels in lesional skin biopsies | Baseline to Week 12

SECONDARY OUTCOMES:
Demonstrate a change in IL-1⍺, IL-23p19, IL-17A, IL-5, IL-6, TNF⍺, HBD-2 protein levels in lesional skin biopsies | Baseline to Week 12
Demonstrate a change in IL-1β, IL-1⍺, IL-23p19, IL-17A, IL-5, IL-6, TNF⍺, HBD-2 mRNA expression in lesional skin biopsies | Baseline to Week 12
Demonstrate a change in IL-1β, IL-1⍺, IL-23p19, IL-17A, IL-5, IL-6, TNF⍺, HBD-2 protein levels in serum | Baseline to Week 12
Demonstrate a change in serum amyloid A levels | Baseline to Week 12
Change in Pain, as measured using a 10-point numerical rating scale, 1 through 10, with 10 being the worst. | Baseline to Week 12
Change in Quality of Life using Dermatology Life Quality Index (DLQI) | Baseline to Week 12
Change in clinical status using the Hurley Staging | Baseline to Week 12
Change in clinical status using the International Hidradenitis Suppurative Severity Score System (IHS4) | Baseline to Week 12
Change in clinical status using the Hidradenitis Suppurative Clinical Response (HiSCR) | Baseline to Week 12
Change in clinical status using the Hidradenitis Suppurative Physician Global Assessment (HS-PGA) | Baseline to Week 12
Change in clinical status using the Hidradenitis Suppurative Area and Severity Index-Revised (HASI-R) | Baseline to Week 12
Change in abscesses and inflammatory nodules count (AN count) | Baseline to Week 12

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Phoenicis Investigative Site, Redwood City, California
  - Phoenicis Investigative Site, Worcester, Massachusetts
  - Phoenicis Investigative Site, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No